CLINICAL TRIAL: NCT06194032
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Four-Way Crossover Phase I Thorough QTc Study to Investigate the Effect on QTcF of Single Doses of Baxdrostat Compared With Placebo, Using Open-label Moxifloxacin as a Positive Control, in Healthy Participants
Brief Title: A Study to Investigate the Effect on QTcF of Baxdrostat Compared With Placebo, Using Moxifloxacin as a Positive Control, in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D6970C00004; 2023-506108-23-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-12-21; First posted 2024-01-08 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Aldosterone synthase inhibitor; QT/QTc interval; Moxifloxacin
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is double-blinded with regard to treatment (baxdrostat or placebo), for all placebo-controlled dose groups (groups where placebo and active substance is given in a cohort, ie, the sponsor, the investigator, all clinical staff involved in the clinical study (except for the unblinded pharmacist), the participants, and the study monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding). Moxifloxacin will be administered as an open-label positive control in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment Sequence ABCD (Experimental): Dummy sequence according to CSP: Participants will receive a single dose of all 4 treatments (ABCD) in a crossover design with a washout period of at least 7 days between each study dose administration.
  Interventions: Drug: Baxdrostat; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence BDAC (Experimental): Dummy sequence according to CSP: Participants will receive a single dose of all 4 treatments (BDAC) in a crossover design with a washout period of at least 7 days between each study dose administration.
  Interventions: Drug: Baxdrostat; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence CADB (Experimental): Dummy sequence according to CSP: Participants will receive a single dose of all 4 treatments (CADB) in a crossover design with a washout period of at least 7 days between each study dose administration.
  Interventions: Drug: Baxdrostat; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence DCBA (Experimental): Dummy sequence according to CSP: Participants will receive a single dose of all 4 treatments (DCBA) in a crossover design with a washout period of at least 7 days between each study dose administration.
  Interventions: Drug: Baxdrostat; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Baxdrostat — Participants will receive baxdrostat as two separate doses.
Drug: Placebo — Participants will receive baxdrostat matching placebo.
Drug: Moxifloxacin — Participants will receive a single dose moxifloxacin

SUMMARY:
This study will assess the effect of single oral doses of baxdrostat on the ECG interval measured from the onset of the QRS complex to the end of the T wave (QT) interval corrected for HR using Fridericia's formula (QTcF) compared to placebo using a concentration-QTcF analysis, and with moxifloxacin as positive control, in healthy participants.

DETAILED DESCRIPTION:
This is a randomised, placebo-controlled, double-blind, 4-way crossover TQT study to assess the effect of single oral doses of baxdrostat on the QTcF compared to placebo using a concentration-QTcF analysis, and with open-label moxifloxacin as positive control, in 28 healthy participants, performed at a single clinical unit.

The study will comprise of:

* a screening period of maximum 28 days,
* four treatment periods during which participants will be resident at the Clinical Unit from Treatment Period Day -1 until at least 48 hours after dosing (Treatment Period Day 3).
* a final Follow-up Visit within 7 to 10 days following discharge after Visit 5

Participants will each receive a single dose of all treatments in a cross-over design over 4 treatment periods. Participants will be randomised to 1 of 4 treatment sequences with equal allocation regarded as a Williams design of order 4.

Treatment Periods will be separated by a washout period of at least 7 days but no more than 9 days.

ELIGIBILITY:
Inclusion Criteria:

* Females must have a negative pregnancy test.
* Have a Basal Metabolic index (BMI) between 19 and 30 kg/m2 inclusive and weigh at least 50 kg.

Exclusion Criteria:

* History of any clinically significant disease or disorder.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of additional risk factors for Torsade de Pointes.
* History of neoplastic disease.
* Family history of sudden cardiac death.
* Any skin condition likely to interfere with ECG electrode placement or adhesion.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of drug.
* Any clinically significant abnormalities at screening and first admission in rhythm, conduction, or morphology of the 12-lead resting ECG and any clinically important abnormalities in the 12-lead ECG as considered by the investigator.
* Participant has clinical signs and symptoms consistent with COVID-19.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
* Positive screen for drugs of abuse, alcohol or cotinine at screening or on each admission to the Clinical Unit.
* Participants who have previously received Baxdrostat.
* Participants with any special dietary restrictions such as participants who are lactose intolerant or are vegetarians/vegans.
* Participants who cannot communicate reliably with the investigator and/or are not able to read, speak, and understand the local language.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Placebo corrected change from baseline in QTcF (ΔΔQTcF) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of single doses of baxdrostat on QTcF compared to placebo using a concentration-QTcF analysis will be assessed.

SECONDARY OUTCOMES:
Heart Rate (HR) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on HR will be assessed.
RR interval | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on RR interval will be assessed.
PR interval | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on PR interval will be assessed.
QRS interval | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on QRS interval will be assessed.
Change from baseline in Heart rate (ΔHR) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on HR will be assessed.
QT interval | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on QT interval will be assessed.
Change from baseline in RR interval (ΔRR) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔRR interval will be assessed.
Change from baseline in PR interval (ΔPR) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔPR interval will be assessed.
Change from baseline in QRS interval (ΔQRS) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔQRS interval will be assessed.
Change from baseline in QTcF (ΔQTcF) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔQTcF will be assessed.
Change from baseline in QT interval (ΔQT) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔQT interval will be assessed.
Number of participants with significant change in QTcF | Day 1 to Day 3
  The presence of categorical outliers for QTcF after baxdrostat administration will be assessed.
Number of participants with significant change in PR interval | Day 1 to Day 3
  The presence of categorical outliers for PR interval after baxdrostat administration will be assessed.
Number of participants with significant change in QRS interval | Day 1 to Day 3
  The presence of categorical outliers for QRS interval after baxdrostat administration will be assessed.
Number of participants with significant change in RR interval | Day 1 to Day 3
  The presence of categorical outliers for RR interval after baxdrostat administration will be assessed.
Number of participants with significant change in QT interval | Day 1 to Day 3
  The presence of categorical outliers for QT interval after baxdrostat administration will be assessed.
Number of participants with significant change in HR | Day 1 to Day 3
  The presence of categorical outliers for HR after baxdrostat administration will be assessed.
Placebo corrected change from baseline in HR (ΔΔHR) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔΔHR will be assessed.
Placebo corrected change from baseline in RR interval (ΔΔRR) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔΔRR interval will be assessed.
Placebo corrected change from baseline in PR interval (ΔΔPR) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔΔPR interval will be assessed.
Placebo corrected change from baseline in QRS (ΔΔQRS) | Visit 2,3, 4 and 5:- Day 1: Pre-dose, 0.5, 1, 1.5, 2,3,4,5,6, 8 and 12 hour (h); Day 2: 24 and 36 h post-dose; Day 3: 48 h post dose
  The effect of baxdrostat on ΔΔQRS interval will be assessed.
AUClast of Baxdrostat | Day 1 to Day 3
  The PK of baxdrostat will be assessed.
AUCinf of Baxdrostat | Day 1 to Day 3
  The PK of baxdrostat will be assessed.
Maximum observed plasma peak concentration (Cmax) of baxdrostat | Day 1 to Day 3
  The PK of baxdrostat will be assessed.
Time to reach peak or maximum observed concentration (Tmax) of baxdrostat | Day 1 to Day 3
  The PK of baxdrostat will be assessed.
Number of participants with Adverse Events (AEs) | Day 1 to last day of follow-up (approximately 7 to 10 days after the last dose)
  The safety and tolerability of baxdrostat will be assessed.
Number of participants with Adverse events of special interest | Day 1 to last day of follow-up (approximately 7 to 10 days after the last dose)
  The safety and tolerability of baxdrostat will be assessed. For this clinical study, AESIs include the following: hyperkalaemia, hyponatraemia, and hypotension events that require intervention.
Number of treatment-emergent changes in T-wave morphology | Day 1 to Day 3
  Morphological changes in the T-wave after baxdrostat administration will be assessed.
Number of treatment-emergent changes in U-waves presence and morphology | Day 1 to Day 3
  Morphological changes in the U wave after baxdrostat administration will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D6970C00004_Redacted_CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6970C00004&attachmentIdentifier=da978a59-c890-4e0a-b691-ca078d43a795&fileName=D6970C00004_Redacted_CSR_Synopsis.pdf&versionIdentifier=
- See also: Results posted on AZCT.com — https://www.astrazenecaclinicaltrials.com/study/D6970C00004/